CLINICAL TRIAL: NCT03404843
Title: Red Blood Cell ATP Release and Vascular Function in Humans
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Colorado State University (Other)
Responsible Party: Principal Investigator, Frank Dinenno, Professor, Colorado State University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 16-6361H
Record Dates: First submitted 2017-11-07; First posted 2018-01-19 (Actual); Results first posted 2020-02-27 (Actual); Last update posted 2020-02-27 (Actual); Status verified 2020-02

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases | interventions — fasudil; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: This is a randomized, double-blind, placebo-controlled, crossover study. Approximately 20 young and 20 older adults will be recruited for participation and randomly assigned to either a placebo (saline) infusion or a fasudil hydrochloride infusion. The dose of fasudil hydrochloride is 60 mg/ 60 min.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: A person not associated with any data collection or data analysis is randomizing the treatment and preparing it in a separate room. All data is collected as visit 1 or visit 2.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Fasudil hydrochloride (Experimental): Participants will receive a 100 mL intravenous infusion (in 60 minutes) of 60 mg of fasudil hydrochloride + saline prior to measurements of vascular function and ATP release.
  Interventions: Drug: Fasudil Hydrochloride
- Saline (Placebo Comparator): Participants will receive a 100 mL intravenous infusion (in 60 minutes) of saline (placebo) prior to measurements of vascular function and ATP release.
  Interventions: Other: Saline

INTERVENTIONS:
Drug: Fasudil Hydrochloride — 10 mg/mL vial of fasudil hydrochloride. 6 mL (60 mg) of fasudil hydrochloride are added to a 100 mL saline bag for delivery to subjects.
  Arms: Fasudil hydrochloride
Other: Saline — 100 mL saline bag.
  Other Names: Placebo
  Arms: Saline

SUMMARY:
Previous work demonstrates that the red blood cells of older adults do not release a potent vasodilator (ATP) as well as the red blood cells of younger adults. The investigators are targeting a pathway within the red blood cell using fasudil hydrochloride to determine if both the release of ATP from red blood cells and blood flow responses to low oxygen (hypoxia) and exercise in older adults can be improved.

DETAILED DESCRIPTION:
Participants will initiate contact with the investigators by responding to flyers placed in the community either by phone or email. The first correspondence (phone or email) will provide a brief description of the research and ask a series of screening questions to determine age, height, weight, and any medications participants may be taking as well as the current health status (diagnoses, basic health history, and physical activity level) of participants. If they qualify, a two hour screening visit is scheduled during a time when the participant will be examined by the physician. All participants will undergo informed consent in a face to face private meeting with the research coordinator. Following informed consent, participants will be evaluated by a physician and undergo a treadmill stress test to rule out cardiovascular disease.

During the study, heart rate will be monitored with a 3-lead ECG and blood pressure will be monitored noninvasively with a blood pressure cuff on the finger (finometry). Venous blood will be collected at multiple time points via a catheter inserted into a forearm vein draining skeletal muscle circulation for measurement of blood gases (0.5 mL/sample) and plasma [ATP] (2 mL/sample), with less than 100 mL of blood being drawn in total (~60mL total). Blood flow at rest and in response to hypoxia and exercise will be measured non-invasively using Doppler ultrasound of the brachial artery. Hypoxia trials will be performed by having participants breathe a low oxygen gas mixture via a mouthpiece that is hooked up to gas tanks and an anesthesia monitor to decrease their oxygen saturation to ~80% (similar to hiking a 14er) for 10 minutes. Exercise trials will last for approximately 15 minutes and will involve participants performing graded-intensity rhythmic handgrip exercise by lifting weights (corresponding to a low, moderate, and high workload) using a pulley system. The drug treatment used in this study (fasudil) is being given because it may improve red blood cell ATP release in older adults. This is a double-blinded placebo controlled study, thus participation will occur on two randomized experimental days.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Sedentary to moderately active
* 18 to 30 years old for young subjects
* 60 to 80 years old for older subjects

Exclusion Criteria:

* Obesity (BMI ≥ 30 kg/m^2)
* Cardiovascular disease
* Metabolic disease
* Use of medications that can influence cardiovascular function
* Blood pressure greater than or equal to 140/90
* Smoker
* Use of hormone replacement therapy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2017-07-14 (Actual); Primary Completion 2018-10-05 (Actual); Study Completion 2018-10-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frank Dinenno, PhD, Principal Investigator — Colorado State University
Locations (1):
- Colorado State University, Dept. of Health and Exercise Science, Fort Collins, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Fasudil, Then Saline: Participants were randomized to receive a single 100 mL intravenous infusion of 60 mg fasudil hydrocholoride + saline in 60 minutes prior to measurements of vascular function and ATP release. After a washout period of at least 5 days, participants received a single 100 mL intravenous infusion of saline (placebo) in 60 minutes prior to measurements of vascular function and ATP release.
- Saline, Then Fasudil: Participants were randomized to receive a single 100 mL intravenous infusion of saline (placebo) in 60 minutes prior to measurements of vascular function and ATP release. After a washout period of at least 5 days, participants received a single 100 mL intravenous infusion of 60 mg fasudil hydrocholoride + saline in 60 minutes prior to measurements of vascular function and ATP release.
Period: Overall Study
Arm/Group | Fasudil, Then Saline | Saline, Then Fasudil
Started | 17 | 14
Completed | 13 | 13
Not Completed | 4 | 1
Not completed — Study difficulties unrelated to Tx | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fasudil, Then Saline | Saline, Then Fasudil | Total
Number analyzed (Participants) | 13 | 13 | 26
Age, Customized [Count of Participants; unit: Participants]
  18-30 years | 6 | 6 | 12
  60-80 years | 7 | 7 | 14
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 13
  Male | 6 | 7 | 13
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 13 | 12 | 25
  Asian | 0 | 1 | 1
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 12 | 12 | 24
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 24.9 (4.0) | 23.7 (1.6) | 24.3 (3.0)

OUTCOME MEASURES:

1. Primary Outcome: Forearm Blood Flow Responses to Hypoxia After Administration of Intervention
Description: Forearm blood flow measured using Doppler ultrasound before and after 5 minutes of exposure to hypoxia (breathing a mix of low-oxygen gas and room air to achieve oxygen saturations of ~80%).
Time Frame: Within 4 hours after administration of intervention
Population: All participants who completed both interventions (crossover design) with outcome data collected
Measure: Mean (Standard Error); unit: mL/min
Groups:
- Young Saline; Older Saline: Participants received a 100 mL intravenous infusion (in 60 minutes) of saline (placebo) prior to outcome measurements
- Young Fasudil; Older Fasudil: Participants received a 100 mL intravenous infusion (in 60 minutes) of 60 mg of fasudil hydrochloride + saline prior to outcome measurements
Arm/Group | Young Saline | Young Fasudil | Older Saline | Older Fasudil
Number analyzed (Participants) | 11 | 11 | 13 | 13
mL/min | 6.3 (1.2) | 6.2 (1.2) | 2.1 (0.6) | 8.4 (1.9)
Statistical Analysis 1: Comparison: Young Saline vs Young Fasudil; Within group comparison of treatment; Test type: Other; p = 0.97, ANOVA
Statistical Analysis 2: Comparison: Older Saline vs Older Fasudil; Within group comparison of treatment; Test type: Other; p < 0.05, ANOVA

2. Primary Outcome: Forearm Blood Flow Responses to Exercise After Administration of Intervention
Description: Forearm blood flow measured using Doppler ultrasound before and during continuous rhythmic handgrip exercise at a low, moderate, and high intensity workload (4 minutes at each workload for 12 minutes in total).
Time Frame: Within 4 hours after administration of intervention
Population: All participants who completed both interventions (crossover design) with outcome data collected
Measure: Mean (Standard Error); unit: mL/min
Arm/Group | Young Saline | Young Fasudil | Older Saline | Older Fasudil
Number analyzed (Participants) | 12 | 12 | 13 | 13
mL/min | 315.4 (31.0) | 283.0 (25.4) | 255.3 (19.9) | 304.2 (25.2)
Statistical Analysis 1: Comparison: Young Saline vs Young Fasudil; Within group comparison of treatment; Test type: Other; p < 0.05, ANOVA
Statistical Analysis 2: Comparison: Older Saline vs Older Fasudil; Within group comparison of treatment; Test type: Other; p < 0.05, ANOVA

3. Primary Outcome: Change in ATP Release to Hypoxia After Administration of Intervention
Description: Venous plasma concentrations of ATP measured using a luminometer before and after 5 minutes of exposure to hypoxia (breathing a mix of low-oxygen gas and room air to achieve oxygen saturations of ~80%).
Time Frame: Within 4 hours after administration of intervention
Population: All participants who completed both interventions (crossover design) with outcome data collected
Measure: Mean (Standard Error); unit: nmol/L
Arm/Group | Young Saline | Young Fasudil | Older Saline | Older Fasudil
Number analyzed (Participants) | 9 | 9 | 11 | 11
nmol/L | 21.6 (10.5) | 5.3 (8.0) | 5.3 (5.4) | 17.4 (13.2)
Statistical Analysis 1: Comparison: Young Saline vs Young Fasudil; Within group comparison of treatment; Test type: Other; p = 0.28, ANOVA
Statistical Analysis 2: Comparison: Older Saline vs Older Fasudil; Within group comparison of treatment; Test type: Other; p = 0.37, ANOVA

4. Primary Outcome: Change in ATP Release to Exercise After Administration of Intervention
Description: Venous plasma concentrations of ATP measured using a luminometer before and during continuous rhythmic handgrip exercise at a low, moderate, and high intensity workload (4 minutes at each workload for 12 minutes in total).
Time Frame: Within 4 hours after administration of intervention
Population: All participants who completed both interventions (crossover design) with outcome data collected
Measure: Mean (Standard Error); unit: nmol/L
Arm/Group | Young Saline | Young Fasudil | Older Saline | Older Fasudil
Number analyzed (Participants) | 12 | 12 | 12 | 12
nmol/L | 45.6 (16.8) | 42.2 (15.1) | 28.4 (7.9) | 46.2 (15.2)
Statistical Analysis 1: Comparison: Young Saline vs Young Fasudil; Within group comparison of treatment; Test type: Other; p = 0.89, ANOVA
Statistical Analysis 2: Comparison: Older Saline vs Older Fasudil; Within group comparison of treatment; Test type: Other; p = 0.30, ANOVA

5. Secondary Outcome: Arterial Stiffness After Administration of Intervention
Description: Arterial stiffness measured non-invasively using a SphygmoCor system after administration of saline (placebo) and fasudil. This is a randomized crossover design study, so participants will receive 1 treatment (saline or fasudil) on their first visit and the other treatment on their second visit.
Time Frame: Immediately following administration of intervention
Population: All participants who completed both interventions (crossover design) with outcome data collected
Measure: Mean (Standard Error); unit: m/s
Arm/Group | Young Saline | Young Fasudil | Older Saline | Older Fasudil
Number analyzed (Participants) | 12 | 12 | 13 | 13
m/s | 5.4 (0.2) | 5.2 (0.2) | 7.8 (0.4) | 7.6 (0.4)
Statistical Analysis 1: Comparison: Young Saline vs Young Fasudil; Within group comparison of treatment; Test type: Other; p = 0.08, ANOVA
Statistical Analysis 2: Comparison: Older Saline vs Older Fasudil; Within group comparison of treatment; Test type: Other; p = 0.05, ANOVA

ADVERSE EVENTS:
Time Frame: During study visits and 1 month after (as reported by participants)
Arm/Group | Young Saline | Young Fasudil | Older Saline | Older Fasudil
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12 | 0/13 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/13 | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2018-05-19): https://cdn.clinicaltrials.gov/large-docs/43/NCT03404843/Prot_000.pdf
  • Statistical Analysis Plan (2018-05-19): https://cdn.clinicaltrials.gov/large-docs/43/NCT03404843/SAP_001.pdf